CLINICAL TRIAL: NCT06170307
Title: Assessment of Left Atrial Function of COVID-19-recovered Patients During the Surge of Omicron Variants by Two-dimensional Speckle Tracking Echocardiography
Brief Title: Left Atrial Function of COVID-19-recovered Patients During the Surge of Omicron Variants
Status: Completed | Type: Observational
Sponsor: Haiyan Wang (Other)
Responsible Party: Sponsor-Investigator, Haiyan Wang, Director, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(136)
Record Dates: First submitted 2023-12-11; First posted 2023-12-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19; Long COVID-19 syndrome; 2-dimensional speckle tracking imaging; echocardiography; Left atrial strain
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COVID-19 group: Patients diagnosed with SARS-CoV-2 Omicron variant infection by SARS-CoV-2 RT-PCR test within 3 months who came to our hospital for echocardiography were included in the case group .
  Interventions: Other: two-dimensional speckle tracking echocardiography
- Control group: Healthy participants were confirmed free of COVID-19 disease by reverse transcriptase-polymerase chain reaction (RT-PCR) testing and computed tomography (CT) imaging.
  Interventions: Other: two-dimensional speckle tracking echocardiography

INTERVENTIONS:
Other: two-dimensional speckle tracking echocardiography — The structural and functional parameters of the left atrial were obtained by conventional echocardiography, and the left atrial strain parameters were obtained by two-dimensional speckle tracking echocardiography.

SUMMARY:
The goal of this observational study is to retrospectively analyze left atrial function in mild to moderate COVID-19-recovered patients. The main questions it aims to answer are:

* Whether left atrial function is involved in patients with mild to moderate COVID-19 after recovery.
* What are the factors that may be associated with persistent heart-related symptoms (including chest pain, chest tightness, palpitations, shortness of breath, or postural tachycardia) in patients with mild to moderate COVID-19 ?

Participants will undergo transthoracic echocardiography to obtain conventional ultrasound parameters, two-dimensional strain parameters will been obtained through software post-processing, and general clinical data and laboratory test results will been obtained.

DETAILED DESCRIPTION:
The included patients who recovered from COVID-19 infection and healthy people underwent transthoracic echocardiography at the First Affiliated Hospital of Shandong First Medical University from December 20, 2022 to January 20, 2023. Routine data and two-dimensional strain parameters of transthoracic echocardiography of the study subjects were obtained:

1. The echocardiographic examination was performed using a Epiq 7C ultrasound machine, and images were acquired with the patient in left lateral decubitus using a 3.5-5 MHz transducer at a depth of 16 cm. ECG was recorded, and 3 consecutive cardiac cycles of each view were recorded during quiet breathing at 50-80 frames/sec. All patients were subjected to conventional transthoracic echocardiography & Speckle tracking echocardiography (STE). All measurements were taken following the American Society of Echocardiography (ASE) recommendations.
2. Left atrial strain analysis was obtained using automated speckle tracking software. The regions of interest were generated automatically and Left atrial endocardial border was manually adjusted when required. Left atrial phases definition and Left atrial strain values were measured from the Left atrial longitudinal strain curve according to the European Association of Cardiovascular Imaging (EACVI)/American society of echocardiography (ASE) guidelines. Global LV systolic strain was evaluated, and the software automatically traced the contour of the endocardium at apical three, four and two-chamber views.
3. At the same time, the general clinical data, demographic characteristics, electrocardiogram, chest CT results, troponin I (hsTnI) and brain natriol peptide levels on the day of echocardiographic examination were obtained through the hospital electronic medical record His system.
4. Clinical follow-up was performed 12-18 months after the echocardiographic examination by phone and by electronic health record review. We recorded: 1) persistent cardiac symptoms, 2) interval presentation to the emergency department or hospitalization with cardiac symptoms, and 3) any major adverse cardiac event (myocardial infarction, stroke, revascularization, or death).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients having been diagnosed with SARS-CoV-2 Omicron variant infection based on real-time reverse-transcription polymerase chain reaction (RT-PCR) results; 2. Asymptomatic or mild to moderate COVID-19 patients. 3.COVID-19 patients who came to our hospital for echocardiography within 3 months after recovery.

Exclusion Criteria:

* Patients with decreased left ventricular ejection fraction (less than 50%), left ventricular segmental wall motion abnormalities, cardiomyopathy, severe valvular heart disease, arrhythmia, thyroid dysfunction, pulmonary hypertension, past or current pulmonary embolism, severe chronic obstructive pulmonary disease, malignancy/renal failure (less than 30) ml/min) or poor cardiogram image quality were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have recovered from mild to moderate COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Left atrial strain | After recruiting, left atrial strain collected through software post-processing analysis will be assessed and reported up to 8 weeks.
  Myocardial strain derived from speckle-tracking echocardiography has been shown to be more sensitive and accurate in detecting subclinical impairment of cardiac function than conventional echocardiography. LV diastolic dysfunction could be explained by Left atrial strain.

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou B, Zhang Y, Han S, Zhang J, Song L, Wang H. Myocardial Dysfunction and Risk of Long COVID in Patients Recovered From Mild and Moderate COVID-19. Echocardiography. 2025 Mar;42(3):e70120. doi: 10.1111/echo.70120. PMID 40029146